CLINICAL TRIAL: NCT04235881
Title: Efficacy of Mindfulness Training on the Quality of Life of Patients With Implantable Automatic Defibrillator
Brief Title: Emotional Regulation in Patients With Implanted Automatic Defibrillator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MF_DAI_La_PAZ
Record Dates: First submitted 2019-11-29; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Arrhythmia; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: Implantable automatic defibrillator; Emotional regulation; MBSR; App; Quality of life; Mindfulness; Anxiety; Depression
MeSH Terms: conditions — Arrhythmias, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular; Emotional Regulation; Alzheimer Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The experimental study was developed through a randomized controlled clinical trial, with simple random probabilistic sampling. With a pre-post design, the variables measured in the participants before performing the mindfulness training were measured again at the end of the program, eight weeks later, in order to compare the values of both measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBSR group (Experimental): Enforcement of the standardized program Mindfulness-Based Stress Reduction
  Interventions: Behavioral: Mindfulness-based stress reduction program
- App group. (Experimental): Enforcement of the emotional regulation program based on mindfulness (ERM) through the mobile phone application REM volver a casa
  Interventions: Behavioral: App REM volver a casa
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction program — Mindfulness training through an adaptation of the standardized MBSR program. This program was conducted in person and in a group, with a maximum of 25 participants per group and a total duration of 8 weeks. The training was carried out in 8 sessions, one each week, with a duration of 2 h each session.
  Arms: MBSR group
Behavioral: App REM volver a casa — The intervention was carried out through the computer application for mobile phone "REM volver a casa". This application has been developed to carry out training in the emotional regulation program based on mindfulness, autonomously. The application is designed to carry out the program in 8 weeks.
  Arms: App group.

SUMMARY:
The general objective of the study was to evaluate the impact of two emotional regulation programs, one standardized and face-to-face (MBSR: Mindfulness Based Stress Reduction) and, another, implemented through a mobile phone application (REM_Volver a casa; ERBM_Back home: Emotional Regulation Based on Mindfulness), on the quality of life, the state emotional and psychological and biological variables associated with stress, in a sample of patients with ICD (implantable cardioverter defibrillator).

The working hypotheses were that after training in emotional regulation, patients with ICD would have better quality of life, lower symptoms of anxiety, depression and hostility, and lower incidence of ventricular arrhythmias than patients in the control group, as well as that there would be no differences between the two tools used for training.

DETAILED DESCRIPTION:
The recruitment process of the participants was carried out by telephone, by the medical staff of the arrhythmia's section, who informed the patients the characteristics and objectives of the study.

The sample size was estimated considering an alpha risk of 0.05 and a beta risk of 0.2, in a bilateral contrast, to detect a difference equal to or greater than 10 units in the Quality of life variable. A standard deviation of 20 points and a 20% loss rate were assumed. The estimated n was 237 patients, to distribute in three branches of 79 patients each.

Before beginning the intervention, participants were informed about the research, and were offered the opportunity to ask questions in order to clarify any doubts about it. Next, they were given a Participant Data Collection Notebook. The Notebook included the information on the investigation and the Informed Consent, to be completed and signed; the request for demographic data (age, gender, educational level, etc.); and, the four questionnaires used to assess the psychological variables of study: SF-36 (quality of life), HADS (anxiety and depression), STAXI (hostility) and FFMQ (Mindfulness) For the descriptive analysis, the number of subjects and the corresponding percentage was used in the qualitative variables. In the quantitative variables the mean and standard deviation were used when the variables adjusted to the normal distribution; otherwise, the median and interquartile range (first and third quartile) were used. The normality test used was the Shapiro-Wilk.

In the hypothesis contrast of the pre-post values, of the variables with distribution adjusted to normal, the Student´s t statistic was used for paired data; For the variables whose distribution did not conform to normal, the Wilcoxon Test was chosen.

For the contrast of inter-group hypothesis (independent samples with distribution not adjusted to normal), the Mann Whitney test was used.

For the statistical analysis of data, the SPSS program, version 20, was used.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years.
* Be a patient of the University Hospital La Paz and have an ICD implanted whose implant was equal to or greater than three months.
* Sufficient knowledge of the Spanish language.
* Have a mobile phone and the ability to handle applications on the phone.
* Availability and sufficient physical conditions to attend mindfulness training in the face-to-face format.

Exclusion Criteria:

* Be over 75 years old.
* Be waiting for a heart transplant or other operation related to cardiac pathology.
* Have previous training in mindfulness, unless it had been done before 5 years and had not been practiced since then.
* Being diagnosed with a serious mental disorder and being in an acute symptomatic period of the disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | In order to assess the change at the Quality of life variable, was measured just before starting the mindfulness training program and, eight weeks later, after finishing it.
  The questionnaire (SF-36: Short Form) uses a Likert scale of 3 or 5 points, with a range of scores from 0 to 100, average of 50 and standard deviation 10.

SECONDARY OUTCOMES:
Anxiety and Depression | In order to assess the change at the anxiety and depression variables, were measured just before starting the mindfulness training program and, eight weeks later, after finishing it.
  HADS: Hospital Anxiety and Depression Scale. This scale assess the presence of anxiety or depression. It consists of two sub-scales, of 7 items each, are scored on a Likert scale of 4 points. The cut-off points used for the two scales were: 0 to 7 = no clinical significance; from 8 to 10 = doubtful; from 11 to 14 = moderate; from 15 to 21 = severe.
Anger | In order to assess the change at the Anger variable, was measured just before starting the mindfulness training program and, eight weeks later, after finishing it.
  STAXI: State-Trait Anger Expression Inventory. Questionnaire used to evaluate the expression of hostility, in terms of personality trait and regarding the circumstantial state at the time of measurement. The scores are represented in standardized T scores: mean of 50 points and a standard deviation of 10 points.
AHR | To assess the change in the AHR variable, the data collected corresponded to the two months before the intervention and the two months after the intervention.
  Average Heart Rate (AHR).These parameters were obtained from the data record of the defibrillator implanted in each patient, and is quantified by beats per minute.
NSVT | To assess the change in the NSVT variable, the data collected corresponded to the two months before the intervention and the two months after the intervention.
  Number of Non-Sustained Ventricular Tachycardia (NSVT). These parameters were obtained from the data record of the defibrillator implanted in each patient, and is quantified by whole numbers.
LVEF | The value of this parameter is recorded at the beginning of the study.
  Left Ventricular Ejection Fraction (LVEF). The ejection fraction is the force with which the left ventricle contracts and is related to the patient's prognosis and its symptomatology. This parameter is classified into four levels, according to the percentage.
  1. Less than 40%: heart failure.
  2. From 40 to 55%: below normal heart function.
  3. From 55 to 70%: normal heart function.
  4. Higher than 75%: can indicate a heart condition.
FC | The value of this parameter is recorded at the beginning of the study.
  Functional Class (FC). The functional class for dyspnea is a classification according to the degree to which patients have the feeling of shortness of breath. The functional classification is determined according to the following four levels:
  1. Without any limitation of physical activity.
  2. Slight limitation of physical activity.
  3. Marked limitation of physical activity.
  4. Inability to carry out any physical activity without symptoms.
Number of Shocks | The estimated period of evaluation is up to 8 years. The events (shocks) accounted are for the period between the date of implantation of the device and the date of the last data collection, approximately 33 months after the start of the study.
  Number of shocks produced by the implantable automatic defibrillator, in each patient. Events (shocks) are determined by their registration in the device (implantable automatic defibrillator). The device has a record in which it stores parameters related to the functioning of the heart and the regulation and control processes performed by the device, among them, the shocks it gives in order to restore a situation of ventricular fibrillation or ventricular arrhythmia. This parameter is quantified by whole numbers.
Daily Activity | To assess the change in the Daily Activity variable, the data collected corresponded to the two months before the intervention and the two months after the intervention.
  Number of daily hours of activity, recorded by the implantable automatic defibrillator device. This parameter is quantified in hours.

OTHER OUTCOMES:
Mindfulness attitude | The data corresponding to the mindfulness attitude measured just before starting the mindfulness training program and, eight weeks later, after finishing it.
  FFMQ: Five Facet Mindfulness Questionnaire. In this questionnaire five factors of mindfulness ability are collected: Observe, from 8 to 40 points; Describe, from 8 to 40 points; Act consciously, from 8 to 40 points; Not judge, from 8 to 40 points; and, Not react, from 7 to 35 points.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodríguez Vega, Doctor, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No